CLINICAL TRIAL: NCT06014905
Title: Pilot/Phase I Study of Feasibility of Acquiring Hyperpolarized Imaging in Patients With Meningioma
Brief Title: Feasibility of Acquiring Hyperpolarized Imaging in Patients With Meningioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Javier Villaneuva-Meyer, MD (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); General Electric (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Javier Villaneuva-Meyer, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23924; NCI-2023-05550 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); 5R21EB030899-02 (NIH); 2P01CA118816-11A1 (NIH); 2P01CA118816-16 (NIH)
Record Dates: First submitted 2023-08-11; First posted 2023-08-28 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperpolarized 13C pyruvate, Magnetic Resonance Imaging (Experimental): Participants will receive a single research MR imaging using HP 13C pyruvate, intravenously injected at a rate of 5 ml/second followed by a 20-ml saline flush at 5 ml/second. Safety monitoring, including vital signs and symptom monitoring will be performed for 30 minutes after dosing is completed, 1 to 3 days after dosing, and up to 30 days post scanning procedure. During the follow-up period, study personnel will obtain clinical data from the participants' medical records.
  Interventions: Drug: Hyperpolarized carbon C 13 pyruvate; Procedure: Magnetic Resonance Image (MRI); Other: Saline

INTERVENTIONS:
Drug: Hyperpolarized carbon C 13 pyruvate — Given Intravenously (IV)
  Other Names: Hyperpolarized 13C-Pyruvate; HP C13 pyruvate
Procedure: Magnetic Resonance Image (MRI) — Imaging procedure
  Other Names: MR
Other: Saline — Given IV
  Other Names: Saline Flush

SUMMARY:
This is a Pilot/Phase I clinical study of hyperpolarized 13C (HP 13C) pyruvate injection that includes the acquisition of magnetic resonance (MR) data performed on participants with meningioma to evaluate metabolism and aid in the non-invasive characterization of aggressive tumor behavior

DETAILED DESCRIPTION:
Primary Objective:

I. To assess the feasibility of hyperpolarized 13C MR imaging as a new and unique tool in the characterization of aggressive tumor behavior in participants with meningioma.

Secondary Objectives:

I. To define the most appropriate parameters for obtaining hyperpolarized 13C data from meningioma patients with a run-in study to optimize spatial and temporal resolution and coverage by detecting signal amplitudes and time dynamics.

II. To measure tumor pyruvate-to-lactate, pyruvate-to-alanine, and pyruvate-to-bicarbonate conversion by 13C pyruvate MR imaging in participants with meningioma planning to undergo surgical resection within 4 weeks, using parameters.

Outline:

Participants will receive a single imaging procedure using HP 13C pyruvate. Participants will then be followed-up for 30 days after completion of the study or until voluntary withdrawal or death.

ELIGIBILITY:
Inclusion Criteria:

1. Known (histopathologically confirmed) or presumed meningioma based on imaging with measurable disease on MRI that shows gadolinium enhancement (at least one cm diameter) intracranially (e.g., not confined to skull base alone).

   a. Thirty of the participants plan to have surgical resection within 4 weeks
2. Participants cannot have contraindication to MRI examinations.
3. Age >=18 years.
4. Have a life expectancy of >12 weeks.
5. Karnofsky Performance Status > 60%.
6. Participants must have adequate renal function (creatinine < 1.5 mg/dL) before imaging. This test must be performed within 60 days prior to hyperpolarized imaging scan.
7. Participants must sign an informed consent indicating that they are aware of the investigational nature of this study.
8. Participants must sign an authorization for the release of their protected health information.

Exclusion Criteria:

1. Has any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the patient's ability to participate in this study or any disease that will obscure toxicity or dangerously impact response to the imaging agent.
2. Uncontrolled blood pressure (Systolic BP≥140 mmHg or diastolic BP ≥>=90 mmHg) despite an optimized regimen of antihypertensive medication.
3. Has a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
4. Participants must not be pregnant or breast feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of Hyperpolarized Imaging scan. Effective contraception (men and women) must be used in participants of child-bearing potential.
5. Participants must be excluded from participating in the study if they are not able to comply with the study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who complete 13C pyruvate MR imaging. | Day of MR imaging (1 day)
  All participants who are enrolled in the study and receive any amount of hyperpolarized 13C pyruvate will be included in the primary outcome analysis. The proportion of participants who complete hyperpolarized 13C pyruvate MR imaging will be reported. If the proportion is greater than 0.7, hyperpolarized 13C MR imaging will be determined to be feasible.

SECONDARY OUTCOMES:
Best Magnetic Resonance (MR) imaging protocol ("measurement") to detect altered pyruvate-to-lactate cell metabolism | Day of MR imaging (1 day)
  Five initial patients will be evaluated to establish the spatial and temporal resolution and coverage that yields the best signal amplitudes and time dynamics for measuring tumor pyruvate-to-lactate will be identified.
Best Magnetic Resonance (MR) imaging protocol ("measurement") to detect altered pyruvate-to-alanine cell metabolism | Day of MR imaging (1 day)
  Five initial patients will be evaluated to establish the spatial, temporal resolution and coverage that yield the best signal amplitudes and time dynamics for measuring tumor pyruvate-to-alanine will be identified.
Best Magnetic Resonance (MR) imaging protocol ("measurement") to detect altered pyruvate-to-bicarbonate cell conversion | Day of MR imaging (1 day)
  Five initial patients will be evaluated to establish the spatial and temporal resolution and coverage that yield the best signal amplitudes and time dynamics for measuring tumor pyruvate-to-bicarbonate conversion will be identified.
Mean of pyruvate-to-lactate | Day of MR imaging (1 day)
  The mean and standard deviations of pyruvate-to-lactate ratio will be reported.
Mean of pyruvate-to-alanine | Day of MR imaging (1 day)
  The mean and standard deviations of pyruvate-to-alanine ratio will be reported.
Mean of pyruvate-to-bicarbonate conversion | Day of MR imaging (1 day)
  The mean and standard deviations of pyruvate-to-bicarbonate conversion rate will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Villanueva-Meyer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No